CLINICAL TRIAL: NCT05345184
Title: Feasibility, Acceptability, and Preliminary Effectiveness of a Cognitive Behavioral Suicide Prevention-focused Intervention Tailored to Adults Diagnosed With Schizophrenia Spectrum Disorders: Aim 2 RCT
Brief Title: Cognitive Behavioral Suicide Prevention for Psychosis: Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lindsay Bornheimer, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00211008; R34MH123609 (NIH)
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Suicide; Psychosis
Keywords: suicide prevention; cognitive behavioral therapy; community mental health
MeSH Terms: conditions — Suicide; Psychotic Disorders; Suicide Prevention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Suicide Prevention for psychosis (treatment group) (Experimental): Cognitive Behavioral Suicide Prevention for psychosis (CBSPp) is a behavioral treatment and will be delivered in 10 weekly individual therapy sessions in addition to standard/current services.
  Interventions: Behavioral: Cognitive Behavioral Suicide Prevention for psychosis (CBSPp)
- Services as Usual (SAU; comparison group) (Active Comparator): Services as usual involve standard and current services that clients are eligible for receiving.
  Interventions: Behavioral: Services as Usual (SAU)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Suicide Prevention for psychosis (CBSPp) — Cognitive and behavioral approach to suicide prevention tailored for individuals with psychosis
  Arms: Cognitive Behavioral Suicide Prevention for psychosis (treatment group)
Behavioral: Services as Usual (SAU) — Standard psychiatric and behavioral services provided at community mental health (e.g., case management, medication management)
  Arms: Services as Usual (SAU; comparison group)

SUMMARY:
Investigators will evaluate the feasibility and preliminary effectiveness of modified Cognitive Behavioral Suicide Prevention for psychosis (CBSPp) in comparison to services-as-usual (SAU) in a randomized controlled trial. Investigators will recruit adult clients receiving services at a community mental health (CMH) setting who have a schizophrenia spectrum disorder and recent suicidal thoughts or behaviors within 3 months of screening (n=60). Client participants will be screened, enrolled and randomized to the CBSPp or SAU group. A 4-wave design will include quantitative assessments at baseline (T1), 1-month after baseline (T2), 3-months after baseline (T3), and 5-months after baseline (T4) with in-depth qualitative interviews at T3 for a random sample of adults in the CBSPp group (n=10). Providers (n=12) will be trained to deliver CBSPp and be assessed from T1-T3 to evaluate the implementation process, including in-depth qualitative interviews at T3.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia Spectrum Disorder
* Suicide ideation and/or attempt within 3 months of screening
* Ability to speak and read in English
* 18 to 65 years of age

Exclusion Criteria:

* Requiring emergency care (e.g. imminent plan to harm self) as determined by trained research staff administering the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Inappropriate for behavioral treatment according to own judgment in consultation with a treating clinician CMH
* Impaired capacity (cognitive capacity)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Calgary Depression Rating Scale (CDRS) change from baseline | 3-months after baseline
  A scale to measure depression, higher scores indicate greater depression
Positive and Negative Syndrome Scale (PANSS) change from baseline | 3-months after baseline
  A scale to measure psychosis symptoms, higher scores indicate greater psychosis
Columbia Suicide Severity Rating Scale (C-SSRS) change from baseline | 3-months after baseline
  A scale to measure suicide thoughts and behavior, higher scores indicate greater suicide thoughts and behavior

SECONDARY OUTCOMES:
Beck Hopelessness Scale change from baseline | 3-months after baseline
  A scale to measure hopelessness, higher scores indicate greater hopelessness
Defeat Scale (D Scale) change from baseline | 3-months after baseline
  A scale to measure defeat, higher scores indicate greater defeat
The Entrapment Scale change from baseline | 3-months after baseline
  A scale to measure entrapment, higher scores indicate greater entrapment
Suicide Stroop Task change from baseline | 3-months after baseline
  A cognitive Stroop tasks to assess information processing, information processing is evaluated in time
Resilience Appraisals Scale (RAS) change from baseline | 3-months after baseline
  A scale to measure appraisals, higher scores indicate stronger resilience appraisals
Suicide Concept Sort Task (SCS) change from baseline | 3-months after baseline
  A cognitive card sorting task to assess schemas, cards are sorted as being closely related to not closely related to suicide as a concept

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Upload to NIMH Data Archive

DOCUMENTS (1):
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT05345184/ICF_000.pdf